CLINICAL TRIAL: NCT07156188
Title: The PAPYRUS Study: Permanent vs. Absorbable Sutures in PrimarY Repair of Umbilical HerniaS: A Multicentre, Single-blind, Non-inferiority, Randomized Controlled Trial
Acronym: PAPYRUS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: North York General Hospital (Other); Royal Victoria Hospital Of Barrie (Unknown); London Health Sciences Centre (Other); University of Alberta (Other)
Responsible Party: Principal Investigator, Rachel Liu Hennessey, Clinical Assistant Professor, University of British Columbia; General Surgeon, Vancouver General Hospital, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H24-03475
Record Dates: First submitted 2025-09-03; First posted 2025-09-05 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Hernia Surgery; Umbilical Hernia Repair
Keywords: Umbilical hernia; Hernia repair surgery; Suture use
MeSH Terms: conditions — Hernia, Umbilical | interventions — Polypropylenes; Polydioxanone

STUDY DESIGN:
Intervention Model Description: The PAPYRUS Trial is the first Canada-wide, multi-centre, prospective, parallel arm, non-inferiority, single blind randomized controlled trial of patients undergoing elective suture repair of small (≤2cm) primary umbilical hernia comparing non-absorbable (polypropylene) suture control group versus absorbable (polydioxanone) suture intervention group. An online web-based central method (built-in on UBC FoM REDCap) will be used for randomization. Randomization must occur intraoperatively to ensure the exclusion criteria that can only be determined during surgery are met and the surgeon confirms defect size. Participants will be followed up at 30 days, 12 months, and 2 years following surgery for assessment. The study visits will be aligned with their standard of care clinic visits.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Permenant Suture (Active Comparator): Repair with permanent 0-0 polypropylene suture.
  Interventions: Other: Permanent Suture
- Absorbable Suture (Active Comparator): Repair with an 0-0 polydioxanone suture
  Interventions: Other: Absorbable

INTERVENTIONS:
Other: Permanent Suture — In both control and intervention groups, an open umbilical hernia repair will be performed based on a standardized surgical technique. Dissection and identification of the fascial defect will be performed in a standardized manner. In the control group, a permanent 0-0 polypropylene suture will be used to close the hernia defect in a transverse or vertical interrupted fashion using either the simple interrupted or the figure-of-eight technique. If the surgeon creates an opening in the umbilical skin or extends the skin incision beyond the paraumbilical incision during the procedure, the participant will be excluded from the study.
  Other Names: Control; polypropylene
  Arms: Permenant Suture
Other: Absorbable — In both control and intervention groups, an open umbilical hernia repair will be performed based on a standardized surgical technique. Dissection and identification of the fascial defect will be performed. An 0-0 polydioxanone suture (PDS) will be used to close the hernia defect in either a transverse or vertical interrupted fashion using either simple interrupted or figure-of-eight technique. If the surgeon creates an opening in the umbilical skin or extends the skin incision beyond the paraumbilical incision during the procedure, the participant will be excluded from the study.
  Other Names: Polydioxanone
  Arms: Absorbable Suture

SUMMARY:
Umbilical hernias can be found in over a quarter of the population and comprise of 15% of hernia repairs performed in Canada. While mesh repair is commonly used for larger hernias, smaller hernia defects are often closed with sutures alone. While non-absorbable sutures may have greater tensile strength, the use of absorbable sutures has been found to reduce the risk for wound infection and improve healing. The objective of this multi-centre, nationwide randomized controlled study is to determine whether there is a difference in hernia recurrence when the repair is completed with absorbable polydioxanone suture versus permanent polypropylene suture. The study will also explore post-operative complications and quality of life. Recruitment will take place over 5 years with follow-up at the 30-day, 12-month and 24-month mark following surgery. The results of this trial will be directly applicable to national and international hernia guidelines and will impact the care of thousands of patients.

DETAILED DESCRIPTION:
Umbilical hernias make up a notable proportion of abdominal wall hernia repairs annually. Up to 25% of the population have asymptomatic umbilical hernias when examined using ultrasound. Recent computed tomography studies have identified umbilical hernia in up to 62% of the population. In Canada in 2019, there were 66,234 hernia surgeries performed. Similarly, there are around 175,000 umbilical hernia repairs per year in the United States.

The European Hernia Society (EHS) guidelines classify umbilical hernias by size as small (0-1cm), medium (more than 1 cm up to 4cm), and large (over 4 cm) based on diameter. Although many hernias are asymptomatic, intra-abdominal contents, such as fat or bowel, can protrude through the defect and result in a surgical emergency. Up to 20% of patients with asymptomatic umbilical hernia will later require elective surgery, and another 4% will require emergency surgery.

The EHS guidelines recommend mesh for all hernia repairs to reduce rate of recurrence, but quality of evidence is limited for hernias less than 1cm in size and therefore suture repair can be considered in these situations. Despite EHS guidelines, in many cases, umbilical hernias up to 2 cm in size are repaired with suture based on intra-operative assessment, for example, to avoid enlarging the defect necessary to accommodate a pre-peritoneal mesh with an overlap of 3cm.

The Americas Hernia Society Quality Collaborative Database found that mesh repairs were used for 82% of umbilical hernias >1cm in diameter and 33% of those ≤1cm in diameter. For the National Health Service in England, 50% of umbilical hernias were repaired with mesh. This has led to the controversial reclassification of small hernias to those <2cm in size. Of small (<2cm) umbilical hernias captured by Herniamed, a hernia registry in Germany, Austria, and Switzerland, suture repair was performed for 76.5% of all cases.

The double-blind multicentre randomized controlled trial by Kauffmann and colleagues. compared suture to mesh repair of primary umbilical hernias and found an 8% recurrence rate following suture repair of umbilical hernias 1-2cm in size.

Based on clinical experience, there does appear to be higher rates of granuloma formation, sinus tract formation, and wound complications following the use of non-absorbable sutures. A systematic review and meta-analysis of techniques for the closure of midline abdominal incisions compared absorbable and non-absorbable suture and identified increased pain and suture sinus formation with the use of non-absorbable suture. Another systematic review comparing slowly absorbable versus non-absorbable suture for laparotomy fascial closure found no difference in hernia rate, but a higher rate of suture sinus formation after using non-absorbable suture. Rat models have also demonstrated that slowly absorbable polydioxanone suture may be preferable to permanent polypropylene suture due to a favourable macrophage response. Two large Danish studies compared non-absorbable, slowly absorbable, and quickly absorbable sutures and found no significant difference in recurrence rates.

There is currently insufficient evidence to recommend a suture type or technique for the suture repair of small umbilical hernias. The PAPYRUS Trial will help guide surgical management and suture decisions for thousands of patients annually in North America.

Common umbilical hernia repair complications include wound infection, pain, or hematoma. Multiple terms exist to describe complications following hernia surgery, and the Ventral Hernia Working Group has endeavoured to standardize this nomenclature by defining surgical site occurrence (SSO) and surgical site occurrences requiring procedural intervention (SSOPI). The PAPYRUS Trial will utilize these metrics as outcome variables because SSO will capture suture complications.

Suture type may play a role in reducing risk of recurrence and post-operative complications following primary suture repair of umbilical hernia. There have been no recent systematic reviews or meta-analyses comparing suture types for umbilical hernia. In the systematic review comparing mesh versus suture for elective repair of umbilical hernia, the studies using slowly absorbable suture may favour suture repair, whereas those using permanent suture may favour mesh repair. The European Hernia Society Guidelines state that there is insufficient clinical literature to determine whether permanent or absorbable suture should be used for the primary open repair of small umbilical hernias. This trial is needed to guide the best practices on the use of suture type when performing suture repair of primary umbilical hernia.

The results of this trial will add to the limited evidence base of the surgical management of umbilical hernias ≤2 cm in size and inform treatment guidelines for suture selection in the management of suture repair for primary umbilical hernia. This trial will guide surgical decisions on preferred suture material for primary umbilical hernia repair based on differences or lack of differences in recurrence, SSO, SSOPI, and patient-reported QoL.

Thus, the research question for this trial is: Does slowly absorbable polydioxanone suture compared to permanent polypropylene suture for primary open repair of small <2 cm umbilical hernias result in non-inferior recurrence, SSO, SSOPI, or QoL at 24 months following surgery?

The primary hypothesis is that slowly absorbable polydioxanone suture will be non-inferior (at a non-inferiority margin of 5%) to permanent polypropylene suture for primary repair of small (≤2cm) umbilical hernias for recurrence at 24 months.

Secondary hypotheses are:

1. Slowly absorbable polydioxanone suture is non-inferior to permanent polypropylene suture for primary repair of small (≤2cm) umbilical hernias for SSO and SSOPI at 24 months post-operatively.

Slowly absorbable polydioxanone suture is non-inferior to permanent polypropylene suture for primary repair of small (≤2cm) umbilical hernias in patient-reported QoL as measured by the HerQLes and the SF-12 surveys at 24 months.

All analyses will be conducted on the intention-to-treat (ITT) population. Continuous data will be expressed as means and standard deviations and analyzed using two-sample t-test. Categorical data will be expressed as contingency tables using counts and percentages and analyzed using Chi-squared test or Fisher's exact test.

Recurrence, SSO, and SSOPI will be analyzed as follows:

* Descriptive statistics using Chi-squared test at 30 days, 12 months and 2 years
* Kaplan-Meier survival analysis at 30 days, 12 months and 2 years
* Log-rank test to compare differences in survival distributions
* Cox proportional hazards model to adjust for covariates and obtain estimates for hazard ratio and 95% confidence interval

HerQLes and SF-12 scores:

• Differences between preoperative and postoperative HerQLes and SF-12 scores at 30 days, 12 months, and 2 years will be first evaluated using repeated measures ANOVA. If significant overall event is detected, then pairwise comparisons using paired t-test at 30 days, 12 months, and 2 years with Bonferroni correction will be conducted.

Subgroup analyses will be conducted to evaluate differences in hernia risk factors and sites. All analyses will be conducted using R Statistical Software (v4.5.0; Vienna, Austria).

ELIGIBILITY:
Inclusion Criteria:

1. Elective surgery for primary umbilical hernia with a defect ≤ 2 cm measured clinically or radiographically
2. Age 19 years or older
3. Patient able to give oral and written informed consent

Exclusion Criteria:

1. Umbilical hernia defect > 2 cm measured clinically, radiologically, or intraoperatively with ruler
2. Multiple defects
3. Incisional hernia: prior hernia in area of operation
4. Recurrent umbilical hernia
5. Epigastric hernia
6. Secondary operation performed simultaneously
7. Pregnancy
8. Infected wounds
9. Acute operation (incarcerated or strangulated hernia)
10. BMI ≥ 35 kg/m^2
11. Ascites or liver cirrhosis
12. Peritoneal dialysis
13. Immunosuppression
14. Connective tissue disorder
15. Patient deemed unfit for primary repair at time of surgery based on surgeon discretion at time of operation (e.g. poor tissue quality or unexpected operative finding)
16. Defect is made in the umbilical skin or skin incision extended beyond paraumbilical incision (e.g. sigma or midline extended incision)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 914 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence | 24 months
  Recurrence will be diagnosed clinically at the time of follow-up. Clinical diagnosis of hernia recurrence will be determined by a standard medical assessment (ie. physical exam). In the event that clinical recurrence is uncertain, a computed tomography scan or ultrasound will be performed while the patient performs a Valsalva maneuver.

SECONDARY OUTCOMES:
SSO | 30 days, 12 months, 24 months
  SSO will be diagnosed according to the Ventral Hernia Working Group definition which includes: surgical site infection, seroma, dehiscence, enterocutaneous fistula, surgical site infection, seroma, wound dehiscence, enterocutaneous fistula, wound cellulitis, non-healing incisional wound, fascial disruption, skin or soft tissue ischemia, skin or soft tissue necrosis, wound serous or purulent drainage, stitch abscess, seroma, hematoma, and infected or exposed mesh.
SSOPI | 30 days, 12 months, 24 months
  Surgical Site Occurrences (SSOs) requiring a procedural intervention, defined as wound opening or debridement, suture excision, or percutaneous drainage
Quality of Life - HerQLes | 30 days, 12 months, 24 months
  The Hernia-Related Quality of Life Survey (HerQLes) is a validated patient-reported outcome measure specific to abdominal wall hernias, verified in a subgroup analysis of patients with small hernias. The HerQLes includes 12 statements related to the abdominal wall. Each of the 12 statements is scored from 1 to 6 (strongly disagree to strongly agree, respectively). Each statement covers a domain relevant to hernia-related QoL, and the scores can be compared for each statement and in aggregate. Summary scores are calculated using the following formula: (120-[(20/12)∗(raw score)]).
Quality of Life - SF-12 | 30 days, 12 months, 24 months
  The 12-item Short Form Survey from the RAND Medical Outcomes Study (SF-12) is a general health status questionnaire, a truncated and validated version of the extensively used 36-item Short Form Survey (SF-36), used to assess baseline health and postoperative recovery. The SF-12 is a self-reported health-related QoL questionnaire comprised of 12 items, including 8 domains of health (physical functioning, role functioning physical, bodily pain, general health, vitality, social functioning, role functioning emotional, and mental health). In accordance with prior hernia research, the results of test items will be normalized and expressed in terms of 2 meta-scores: Physical Component Summary and Mental Component Summary. A higher SF-12 score is indicative of better functioning.
Post-Operative Complications | 30 days
  Complications will be determined at follow-up 30 days after surgery and will be defined based on Clavien-Dindo criteria (Clavien et al., 2009).

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - Royal Alexandra Hospital/University of Alberta, Edmonton, Alberta
  - Royal Victoria Hospital, Barrie, Ontario
  - London Health Sciences Centre, London, Ontario
  - North York General Hospital, North York, Ontario
  - Vancouver Coastal Health, Vancouver

IPD SHARING:
Plan to Share IPD: No
Patients will be assigned a unique study ID and no identifiers will be retained for analysis. A master list linking patients' PHN and the study ID will be retained only during data collection to avoid duplication of data entry. The master list will be stored as a password protected Excel spreadsheet on the institutional share drive. Only study personnel will have access to the spreadsheet. Once the collection is completed, this master list will be deleted and data will be completely de-identified. All de-identified data are recorded and stored on each institution's REDCap. Only the Lead Site research team will have the ability to see the entire dataset when processing and analyzing; each collaborating site will only be able to see data they input from their own site. This is to protect patient data, in accordance with provincial health information policies.

REFERENCES:
- [Background] Wright D, Paterson C, Scott N, Hair A, O'Dwyer PJ. Five-year follow-up of patients undergoing laparoscopic or open groin hernia repair: a randomized controlled trial. Ann Surg. 2002 Mar;235(3):333-7. doi: 10.1097/00000658-200203000-00004. PMID 11882754
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Ventral Hernia Working Group; Breuing K, Butler CE, Ferzoco S, Franz M, Hultman CS, Kilbridge JF, Rosen M, Silverman RP, Vargo D. Incisional ventral hernias: review of the literature and recommendations regarding the grading and technique of repair. Surgery. 2010 Sep;148(3):544-58. doi: 10.1016/j.surg.2010.01.008. Epub 2010 Mar 20. PMID 20304452
- [Background] Venclauskas L, Jokubauskas M, Zilinskas J, Zviniene K, Kiudelis M. Long-term follow-up results of umbilical hernia repair. Wideochir Inne Tech Maloinwazyjne. 2017 Dec;12(4):350-356. doi: 10.5114/wiitm.2017.70327. Epub 2017 Sep 26. PMID 29362649
- [Background] van Veen RN, Wijsmuller AR, Vrijland WW, Hop WC, Lange JF, Jeekel J. Randomized clinical trial of mesh versus non-mesh primary inguinal hernia repair: long-term chronic pain at 10 years. Surgery. 2007 Nov;142(5):695-8. doi: 10.1016/j.surg.2007.05.019. PMID 17981189
- [Background] Sajid MS, Parampalli U, Baig MK, McFall MR. A systematic review on the effectiveness of slowly-absorbable versus non-absorbable sutures for abdominal fascial closure following laparotomy. Int J Surg. 2011;9(8):615-25. doi: 10.1016/j.ijsu.2011.09.006. Epub 2011 Oct 30. PMID 22061310
- [Background] Rutkow IM. Demographic and socioeconomic aspects of hernia repair in the United States in 2003. Surg Clin North Am. 2003 Oct;83(5):1045-51, v-vi. doi: 10.1016/S0039-6109(03)00132-4. PMID 14533902
- [Background] Renshaw SM, Gupta A, Poulose BK. Establishing the minimal clinically important difference for the Hernia-Related Quality of Life Survey (HerQLes). Am J Surg. 2022 Feb;223(2):245-249. doi: 10.1016/j.amjsurg.2021.06.018. Epub 2021 Jul 2. PMID 34256930
- [Background] Pawlak M, Tulloh B, de Beaux A. Current trends in hernia surgery in NHS England. Ann R Coll Surg Engl. 2020 Jan;102(1):25-27. doi: 10.1308/rcsann.2019.0118. Epub 2019 Aug 16. PMID 31418302
- [Background] Muysoms F, Campanelli G, Champault GG, DeBeaux AC, Dietz UA, Jeekel J, Klinge U, Kockerling F, Mandala V, Montgomery A, Morales Conde S, Puppe F, Simmermacher RK, Smietanski M, Miserez M. EuraHS: the development of an international online platform for registration and outcome measurement of ventral abdominal wall hernia repair. Hernia. 2012 Jun;16(3):239-50. doi: 10.1007/s10029-012-0912-7. Epub 2012 Apr 18. PMID 22527930
- [Background] Melkemichel M, Bringman S, Granasen G, Widhe B. SUMMER Trial: mesh versus suture repair in small umbilical hernias in adults-a study protocol for a prospective randomized double-blind multicenter clinical trial. Trials. 2021 Jun 22;22(1):411. doi: 10.1186/s13063-021-05366-7. PMID 34158088
- [Background] LaGuardia JS, Milek D, Lebens RS, Chen DR, Moghadam S, Loria A, Langstein HN, Fleming FJ, Leckenby JI. A Scoping Review of Quality-of-Life Assessments Employed in Abdominal Wall Reconstruction. J Surg Res. 2024 Mar;295:240-252. doi: 10.1016/j.jss.2023.10.013. Epub 2023 Dec 2. PMID 38041903
- [Background] Krpata DM, Schmotzer BJ, Flocke S, Jin J, Blatnik JA, Ermlich B, Novitsky YW, Rosen MJ. Design and initial implementation of HerQLes: a hernia-related quality-of-life survey to assess abdominal wall function. J Am Coll Surg. 2012 Nov;215(5):635-42. doi: 10.1016/j.jamcollsurg.2012.06.412. Epub 2012 Aug 4. PMID 22867715
- [Background] Koebe S, Greenberg J, Huang LC, Phillips S, Lidor A, Funk L, Shada A. Current practice patterns for initial umbilical hernia repair in the United States. Hernia. 2021 Jun;25(3):563-570. doi: 10.1007/s10029-020-02164-z. Epub 2020 Mar 11. PMID 32162111
- [Background] Kockerling F, Brunner W, Fortelny R, Mayer F, Adolf D, Niebuhr H, Lorenz R, Reinpold W, Zarras K, Weyhe D. Treatment of small (< 2 cm) umbilical hernias: guidelines and current trends from the Herniamed Registry. Hernia. 2021 Jun;25(3):605-617. doi: 10.1007/s10029-020-02345-w. Epub 2020 Nov 25. PMID 33237505
- [Background] Holihan JL, Flores-Gonzalez JR, Mo J, Ko TC, Kao LS, Liang MK. A Prospective Assessment of Clinical and Patient-Reported Outcomes of Initial Non-Operative Management of Ventral Hernias. World J Surg. 2017 May;41(5):1267-1273. doi: 10.1007/s00268-016-3859-5. PMID 28050665
- [Background] Dias Rasador AC, da Silveira CAB, Lima DL, Nogueira R, Malcher F, Sreeramoju P, Cavazzola LT. Mesh versus suture for elective primary umbilical hernia open repair: a systematic review and meta-analysis. Hernia. 2024 Dec;28(6):2069-2078. doi: 10.1007/s10029-024-03106-9. Epub 2024 Jul 13. Erratum In: Hernia. 2024 Dec;28(6):2445. doi: 10.1007/s10029-024-03175-w. PMID 39001938
- [Background] DeBord J, Novitsky Y, Fitzgibbons R, Miserez M, Montgomery A. SSI, SSO, SSE, SSOPI: the elusive language of complications in hernia surgery. Hernia. 2018 Oct;22(5):737-738. doi: 10.1007/s10029-018-1813-1. Epub 2018 Sep 10. No abstract available. PMID 30203373
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Christoffersen MW, Helgstrand F, Rosenberg J, Kehlet H, Strandfelt P, Bisgaard T. Long-term recurrence and chronic pain after repair for small umbilical or epigastric hernias: a regional cohort study. Am J Surg. 2015 Apr;209(4):725-32. doi: 10.1016/j.amjsurg.2014.05.021. Epub 2014 Jul 31. PMID 25172168
- [Background] Christoffersen MW, Helgstrand F, Rosenberg J, Kehlet H, Bisgaard T. Lower reoperation rate for recurrence after mesh versus sutured elective repair in small umbilical and epigastric hernias. A nationwide register study. World J Surg. 2013 Nov;37(11):2548-52. doi: 10.1007/s00268-013-2160-0. PMID 23887595
- [Background] Bedewi MA, El-Sharkawy MS, Al Boukai AA, Al-Nakshabandi N. Prevalence of adult paraumbilical hernia. Assessment by high-resolution sonography: a hospital-based study. Hernia. 2012 Feb;16(1):59-62. doi: 10.1007/s10029-011-0863-4. Epub 2011 Jul 28. PMID 21796449
- [Background] Antonescu I, Scott S, Tran TT, Mayo NE, Feldman LS. Measuring postoperative recovery: what are clinically meaningful differences? Surgery. 2014 Aug;156(2):319-27. doi: 10.1016/j.surg.2014.03.005. Epub 2014 Mar 15. PMID 24947644
- [Background] Alvarez-Lozada LA, Arrambide-Garza FJ, Quiroga-Garza A, Huerta-Sanchez MC, Escobar-Luna A, Sada-Trevino MA, Ramos-Proano CE, Elizondo-Omana RE. Underdiagnosis of umbilical hernias in CT scans in a multicenter study - the radiologically neglected pathology and its surgical implications. Hernia. 2024 Oct;28(5):1775-1781. doi: 10.1007/s10029-024-03079-9. Epub 2024 Jun 5. PMID 38837076
- [Background] van Steensel S, van den Hil LCL, Bloemen A, Gijbels MJ, Breukink SO, Melenhorst J, Lenaerts K, Bouvy ND. Prevention of incisional hernia using different suture materials for closing the abdominal wall: a comparison of PDS, Vicryl and Prolene in a rat model. Hernia. 2020 Feb;24(1):67-78. doi: 10.1007/s10029-019-01941-9. Epub 2019 May 20. PMID 31111322
- [Background] Kaufmann R, Halm JA, Eker HH, Klitsie PJ, Nieuwenhuizen J, van Geldere D, Simons MP, van der Harst E, van 't Riet M, van der Holt B, Kleinrensink GJ, Jeekel J, Lange JF. Mesh versus suture repair of umbilical hernia in adults: a randomised, double-blind, controlled, multicentre trial. Lancet. 2018 Mar 3;391(10123):860-869. doi: 10.1016/S0140-6736(18)30298-8. Epub 2018 Feb 17. PMID 29459021
- [Background] Henriksen NA, Montgomery A, Kaufmann R, Berrevoet F, East B, Fischer J, Hope W, Klassen D, Lorenz R, Renard Y, Garcia Urena MA, Simons MP; European and Americas Hernia Societies (EHS and AHS). Guidelines for treatment of umbilical and epigastric hernias from the European Hernia Society and Americas Hernia Society. Br J Surg. 2020 Feb;107(3):171-190. doi: 10.1002/bjs.11489. Epub 2020 Jan 9. PMID 31916607
- [Background] Haisley KR, Vadlamudi C, Gupta A, Collins CE, Renshaw SM, Poulose BK. Greatest Quality of Life Improvement in Patients With Large Ventral Hernias: An Individual Assessment of Items in the HerQLes Survey. J Surg Res. 2021 Dec;268:337-346. doi: 10.1016/j.jss.2021.06.075. Epub 2021 Aug 13. PMID 34399356
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Brazier JE, Harper R, Jones NM, O'Cathain A, Thomas KJ, Usherwood T, Westlake L. Validating the SF-36 health survey questionnaire: new outcome measure for primary care. BMJ. 1992 Jul 18;305(6846):160-4. doi: 10.1136/bmj.305.6846.160. PMID 1285753
- [Background] Bergstrom M, Widhe B, Granasen G, Lof Granstrom A, Ohlsson J, Schult S, Dahlstrand U, Osterberg J, Loogna P, Bringman S, Melkemichel M. Onlay mesh versus suture repair for smaller umbilical hernias in adults-early results from SUMMER trial: randomized clinical trial. BJS Open. 2024 Dec 30;9(1):zrae173. doi: 10.1093/bjsopen/zrae173. PMID 40037347
- [Background] Baucom RB, Ousley J, Oyefule OO, Stewart MK, Phillips SE, Browman KK, Sharp KW, Holzman MD, Poulose BK. Evaluation of long-term surgical site occurrences in ventral hernia repair: implications of preoperative site independent MRSA infection. Hernia. 2016 Oct;20(5):701-10. doi: 10.1007/s10029-016-1523-5. Epub 2016 Aug 8. PMID 27502493